CLINICAL TRIAL: NCT06470828
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TAK-861 for the Treatment of Narcolepsy With Cataplexy (Narcolepsy Type 1)
Brief Title: A Study of TAK-861 for the Treatment of Narcolepsy Type 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-861-3001; 2023-508465-32-00 (EU CTIS Number); jRCT2051240083 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Narcolepsy Type 1
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TAK-861 Dose 1 (Experimental): Participants will receive TAK-861 tablets at dose 1, orally, for 12 weeks.
  Interventions: Drug: TAK-861
- TAK-861 Dose 2 (Experimental): Participants will receive TAK-861 tablets at dose 2, orally, for 12 weeks.
  Interventions: Drug: TAK-861
- Placebo (Placebo Comparator): Participants will receive TAK-861-matching placebo tablets, orally, for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-861 — Oral tablet.
  Arms: TAK-861 Dose 1; TAK-861 Dose 2
Drug: Placebo — TAK-861-matching placebo tablet.
  Arms: Placebo

SUMMARY:
The main aim of this study is to learn how effective TAK-861 is in improving excessive sleepiness during the day (called excessive daytime sleepiness or EDS) after 3 months of treatment. Other aims are to learn how effective TAK-861 is in lowering the number of sudden, unexpected attacks of muscle weakness while staying conscious (cataplexy) in a week; to learn the effect TAK-861 has on participants' ability to maintain attention, participant's overall quality of life, the spectrum of narcolepsy symptoms, and daily life functions; and to learn about the safety of TAK-861.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-861. TAK-861 is being tested to evaluate its efficacy and safety in people with narcolepsy type 1 (NT1).

The study will enroll approximately 152 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the three treatment groups:

1. TAK-861 Dose 1
2. TAK-861 Dose 2
3. Placebo

The study drug will be administered for 12 weeks. This multi-center trial will be conducted globally.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has a body mass index (BMI) within the range 18 to 40 kilograms per meter square (kg/m^2).
2. The participant has an International Classification of Sleep Disorders, Third Edition (ICSD-3) or International Classification of Sleep Disorders, Third Edition, Text Revision (ICSD-3-TR) diagnosis of NT1.
3. The participant has greater than or equal to (≥)4 partial or complete episodes of cataplexy/week (WCR).
4. The participant is positive for the human leukocyte antigen (HLA) genotype HLA-DQB1*06:02 or results from radioimmunoassay indicate the participant's cerebrospinal fluid (CSF) orexin (OX)/hypocretin-1 concentration is less than or equal to (≤)110 picograms per milliliter (pg/mL) [or less than one-third of the mean values obtained in normal participants within the same standardized assay].

Exclusion Criteria:

1. The participant has a current medical disorder, other than narcolepsy with cataplexy, associated with EDS.
2. The participant: (a) has a history of myocardial infarction; (b) has a history of clinically significant hepatic disease, thyroid disease, coronary artery disease, cardiac rhythm abnormality or heart failure; or (c) has any medical condition (such as unstable cardiovascular, pulmonary, renal or gastrointestinal disease).
3. The participant has current or recent (within 6 months) gastrointestinal disease that is expected to influence the absorption of drugs.
4. The participant has a history of cancer in the past 5 years.
5. The participant has a clinically significant history of head injury or head trauma.
6. The participant has a history of epilepsy, seizure, or convulsion.
7. The participant has a history of cerebral ischemia, transient ischemic attack (<5 years from screening), intracranial aneurysm, or arteriovenous malformation.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Change From Baseline to Week 12 in Mean Sleep Latency From the 4 Maintenance of Wakefulness Test (MWT) Wake Trials | Baseline, Week 12
  The MWT evaluates a person's ability to remain awake under soporific conditions for a defined period of time. Because there is no biological measure of wakefulness, wakefulness is measured indirectly by the inability or delayed tendency to fall asleep. This tendency to fall asleep is measured via electroencephalography-derived sleep latency in the MWT. The MWT consists of four 40-minute sessions (trials) done 2 hours apart. Sleep latency in each session will be recorded. Participants will be required to stay awake in between the 4 sessions.

SECONDARY OUTCOMES:
Change From Baseline to Week 12 in ESS Total Score | Baseline, Week 12
  The ESS provides individuals with 8 different situations of daily life and asks them how likely they are to fall asleep in those situations (scored 0 to 3) and to try to imagine their likelihood of dozing even if they have not actually been in the identical situation; the scores are summed to give an overall score of 0 to 24. Higher scores indicate stronger subjective daytime sleepiness, and scores below 10 are considered to be within the normal range.
Weekly Cataplexy Rate (WCR) at Week 12 | Week 12
Change From Baseline to Week 12 in Mean Number of Lapses on the 3 Psychomotor Vigilance Test (PVT) | Baseline, Week 12
  The PVT is a simple reaction performance task that aims to measure sustained attention. The change from baseline in the mean number of lapses (delayed responses to a visual cue from intraday sessions) during the 10 minute test will be used as a measure of objective sustained attention.
Patient Global Impression of Change (PGI-C) Score at Week 12 | Week 12
  The PGI-C is a patient self-rated scale to assess improvement in daytime sleepiness and overall narcolepsy symptoms. The PGI-C includes 7 items being scored from 1 (best outcome) to 7 (worst outcome) with 4 being no change.
Change From Baseline to Week 12 in Narcolepsy Severity Scale for Clinical Trials (NSS-CT) Total Score | Baseline, Week 12
  The NSS-CT is a 15-item self-administered questionnaire that assesses the severity and consequences of the 5 major narcolepsy symptoms such as daytime sleepiness, cataplexy, hallucinations, sleep paralysis, and disturbed nighttime sleep (DNS) with a total score range of 0 to 57 (sum of 6 items that assess symptoms severity are rated using a six-point Likert scale [0-5] and 9 items that describe the symptom effect on daily life are rated using a four-point Likert scale [0-3]). Higher total scores mean a worse outcome.
Change From Baseline to Week 12 in Functional Impacts of Narcolepsy Instrument (FINI) Domain Scores | Baseline, Week 12
  The FINI measures the functional impacts of narcolepsy across 6 domains. Each domain is scored from 0 to 4, where 0 indicates the best health and 4 the worst.
Change From Baseline to Week 12 in Short Form-36 Survey (SF-36) Mental and Physical Component Scores | Baseline, Week 12
  The SF-36 is participant-reported survey of participant health that assesses the quality of life and includes both physical and mental components. The scores for each component range from 0 to 100. Higher scores represent better health-related quality of life.
Number of Participants with At Least one Treatment-Emergent Adverse Event (TEAE) | Up to 16 weeks
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product. A TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a study intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the study intervention or medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (53):
- United States (15):
  - Takeda Site 48, Phoenix, Arizona
  - Takeda Site 39, Redwood City, California
  - Takeda Site 31, Santa Ana, California
  - Takeda Site 18, Upland, California
  - Takeda Site 4, Orlando, Florida
  - Takeda Site 3, Atlanta, Georgia
  - Takeda Site 45, Boston, Massachusetts
  - Takeda Site 5, St Louis, Missouri
  - Takeda Site 2, Denver, North Carolina
  - Takeda Site 6, Cincinnati, Ohio
  - Takeda Site 42, Cleveland, Ohio
  - Takeda Site 49, Danville, Pennsylvania
  - Takeda Site 1, Columbia, South Carolina
  - Takeda Site 44, Dallas, Texas
  - Takeda Site 10, Norfolk, Virginia
- Canada (3):
  - Takeda Site 21, Ottawa, Ontario
  - Takeda Site 11, Toronto, Ontario
  - Takeda Site 50, Montreal, Quebec
- France (4):
  - Takeda Site 25, Montpellier, Herault
  - Takeda Site 43, Toulouse, Midi-Pyrenees
  - Takeda Site 40, Lyon
  - Takeda Site 29, Paris
- Germany (3):
  - Takeda Site 47, Regensberg, Bavaria
  - Takeda Site 34, Berlin
  - Takeda Site 26, Schwerin
- Italy (2):
  - Takeda Site 32, Rome, Lazio
  - Takeda Site 30, Bologna
- Japan (11):
  - Takeda Site 16, Kurume-shi, Fukuka-Ken
  - Takeda Site 13, Kitakyushu-shi, Fukuoka
  - Takeda Site 14, Fukuoka, Fukuoka-Shi Hakata-Ku
  - Takeda Site 9, Kohoku, Kanagawa
  - Takeda Site 7, Kumamoto, Kumamoto
  - Takeda Site 17, Isahaya-shi, Nagasaki
  - Takeda Site 15, Urasoe-Shi, Okinawa
  - Takeda Site 12, Yodogawa, Osaka
  - Takeda Site 8, Bunkyo-ku, Tokyo
  - Takeda Site 19, Kodaira-shi, Tokyo
  - Takeda Site 20, Shibuya-ku, Tokyo
- Takeda Site 28, Zwolle, Netherlands
- Norway (2):
  - Takeda Site 27, Bergen, Hordaland
  - Takeda Site 33, Oslo
- Spain (6):
  - Takeda Site 37, Vitoria-Gasteiz, Alava
  - Takeda Site 38, Castellon, Castellon
  - Takeda Site 35, Barcelona
  - Takeda Site 36, Barcelona
  - Takeda Site 24, Madrid
  - Takeda Site 41, Valencia
- Switzerland (3):
  - Takeda Site 22, Barmelweid, Canton of Aargau
  - Takeda Site 23, Bern
  - Takeda Site 51, Lugano
- United Kingdom (3):
  - Takeda Site 46, Cambridge
  - Takeda Site 52, London
  - Takeda Site 53, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/7c9baa5c098c4dcc??page=1&idFilter=TAK-861-3001